CLINICAL TRIAL: NCT05842733
Title: A Novel, Potent and Non-addictive Analgesic of Combinations for Knee Replacement Moderate to Severe Pain Management
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sinew Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oral SDE+AAP-001
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative
Keywords: SafeTynadol; Naldebain
MeSH Terms: conditions — Pain, Postoperative | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Naldebain (Active Comparator): Oral Placebo A 650 mg + Naldebain 37.5 mg (0.5 mL oil solution) + Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.
  Interventions: Drug: Naldebain
- SafeTynadol (Active Comparator): Oral SafeTynadol 650 mg + Placebo B (0.5 mL oil solution) +Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.
  Interventions: Drug: SafeTynadol
- Naldebain + SafeTynadol (Active Comparator): Oral Naldebain 37.5 mg (0.5 mL oil solution) + SafeTynadol 650 mg + Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 25 hours after the first dose.
  Interventions: Drug: Naldebain + SafeTynadol

INTERVENTIONS:
Drug: Naldebain — Oral Placebo A 650 mg + Naldebain 37.5 mg (0.5 mL oil solution) + Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.
  Other Names: Placebo A + Tween20 and PEG400
  Arms: Naldebain
Drug: SafeTynadol — Oral SafeTynadol 650 mg + Placebo B (0.5 mL oil solution) +Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.
  Other Names: Placebo B + Tween20 and PEG400
  Arms: SafeTynadol
Drug: Naldebain + SafeTynadol — Oral Naldebain 37.5 mg (0.5 mL oil solution) + SafeTynadol 650 mg + Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.
  Other Names: Tween20 and PEG400
  Arms: Naldebain + SafeTynadol

SUMMARY:
To assess the safety, efficacy, and pharmacokinetics of oral SafeTynadol, Naldebain and Naldebain combine with SafeTynadol in the treatment of moderate to severe pain following knee replacement.

DETAILED DESCRIPTION:
Randomized, double-blind, parallel-group, 3-arm, oral Placebo A 650 mg + Naldebain 37.5 mg (0.5 mL oil solution) + Tween 20 and PEG 400 (1 capsule), oral SafeTynadol 650 mg + Placebo B (0.5 mL oil solution) + Tween 20 and PEG 400 (1 capsule), oral Naldebain 37.5 mg (0.5 mL oil solution) + SafeTynadol 650 mg + Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.

The complete evaluable 36 subjects (12 subjects in each group) will be analysis in this study. The experiment is divided into three groups of 12 people each. All subjects will be evaluated pharmacokinetics by drawing blood single point at 70.75 ± 2 hours after the first dose..

The population for this study in patients scheduled for knee replacement.

Each group of 12 subjects are administered group 1-3 from day 1-4 after surgery. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose. Mode of administration of oral Naldebain 37.5 mg (0.5 mL oil solution) or Placebo B (0.5 mL oil solution) is withdrawing 0.5 mL of Naldebain 37.5 mg (0.5 mL oil solution) or Placebo B (0.5 mL oil solution) from the vial by a syringe, then is injected into the empty capsule and dispense within 10 minutes prior to dosing.

Screening (Days -30 to -1) (All Study Subjects)

The nature of the study as well as the potential risks and benefits associated with study participation will be fully explained to all potential subjects. The following will then be obtained:

1. Informed consent.
2. Demographic information, including height and weight.
3. Vital signs (temperature, respiratory rate, blood pressure and heart rate).
4. Medical history, including medication use.
5. Complete physical examination including 12-lead ECG.
6. Laboratory testing (blood 50 ± 5 mL) to include the following:

   1. CBC with differential, platelets, White blood cell count (WBC), Red blood cell count (RBC), Hemoglobin, Hematocrit, Mean cell volume (MCV), Mean cell hemoglobin (MCH), Mean cell hemoglobin concentration (MCHC), Platelet count, Differential white cell count.
   2. Blood chemistry screen (Glucose, AST, ALT, BUN, creatinine, K, Na, Antibody screening, ABO Grouping & RH Type, Activated partial thromboplastin time, Prothrombin time).
   3. Galactose single-point (GSP) test.
   4. Urine pregnancy test (female only) (not applicable to female who has stopped menstruating for at least five years).
7. CHEST PA VIEW

Study Day -1

Subjects will be required to check into the clinical site before surgery (Day -1). The following procedures will be performed:

1. Physical examination.*
2. Vital signs.*
3. Urine pregnancy test (female only) (not applicable to female who has stopped menstruating for at least five years).*
4. Review of concomitant medications.*
5. Blood (8 ± 3 mL) will be obtained to assess SDE, nalbuphine, AAP and metabolites (AAP-Sul, AAP-Glc, AAP-Cys, AAP-Nac and APAP-protein adducts) concentrations.

   * If the screening test items are performed in Day -1, the repeat test items only need to be tested once.

Study Day 1-4

All subjects will be given regional anesthesia and be preferentially randomized into one of group 1-3. The study drug will be administered 1-4 days after surgery. First dose of study medication is given 2 ± 2 hours after surgery. Total trial drug will be giving eight times. Each group of 12 subjects are administered group 1-3 from day 1-4 after surgery.

Group 1: Oral Placebo A 650 mg + Naldebain 37.5 mg (0.5 mL oil solution) + Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.

Group 2: Oral SafeTynadol 650 mg + Placebo B (0.5 mL oil solution) +Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 25, 58 ± 2 and 70 ± 2 hours after the first dose.

Group 3: Oral Naldebain 37.5 mg (0.5 mL oil solution) + SafeTynadol 650 mg + Tween 20 and PEG 400 (1 capsule), multiple doses for 3 days. Dosing at 0（2 ± 2 hour after surgery）, 6 ± 2, 14 ± 2, 22 ± 2, 34 ± 2, 46 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.

After surgery, the following evaluations will be performed.

1. Pain assessment: All subjects will assess their average pain intensity using a VAS pain scale. The VAS pain scale assessment will start at 0 ± 0.5, 2 ± 0.5, 4 ± 0.5, 6 ± 2, 10 ± 25, 14 ± 2, 22 ± 2, 28 ± 2, 34 ± 2, 46 ± 2, 52 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.
2. Blood draw (5 ± 3 mL) for assessment of liver chemistry tests (ALT and AST) at 1 ± 0.5 hours after the first oral administration. If significant hepatotoxicity occurs (ALT or AST level more than 5 folds of ULN (upper limit of normal); or ALT or AST level more than 3 folds of ULN with signs of hepatitis, such as jaundice; or ALT or AST > 1000IU), subject needs to withdraw.
3. VAS score assessed for three times in 5-minut e intervals before giving rescue medication. The VAS score is greater than 7 at least two times. VAS score assessed before giving rescue medication as VAS score for the remaining assessments.
4. When the subject takes the study medication or rescue medication, and request further rescue medication. VAS score assessed for three times in 5-minute intervals before giving rescue medication. The VAS score has to greater than 7 at least two times. Rescue medication will be given in the order of (1) to (2). The interval between rescue medications should be at least 1 hour.
5. If the subject requests rescue medicine, the group 1-3 will receive sequence of rescue medications follow the (1) IV Parecoxib 40 mg Q12H and (2) IV morphine 4 mg Q4H PRN.The above method of administration shall be carried out according to the procedure of administration in the hospital ward.
6. Recorded the first time to IV Parecoxib 40 mg and IV morphine 4 mg, and then the amount and frequency of the medications' use within 72 hours will be recorded.
7. Blood draw (8 ± 3 mL) for assessment of SDE, nalbuphine, acetaminophen and metabolites (AAP-Sul, AAP-Glc, AAP-Cys, AAP-Nac and APAP-protein adducts) concentrations before giving the first time's rescue medicationor termination or withdrawals.
8. Vital signs (temperature, respiratory rate, blood pressure and heart rate) will be checked at 0 ± 0.5, 2 ± 0.5, 4 ± 0.5, 6 ± 2, 10 ± 2, 14 ± 2, 22 ± 2, 28 ± 2, 34 ± 25, 46 ± 2, 52 ± 2, 58 ± 2 and 70 ± 2 hours after the first dose.
9. The evaluation of adverse events will continue until the end of the trial 120 hours after the first dose.
10. Review of concomitant medications.
11. Using Brief Pain Inventory short form (BPIsf) to assess pain intensity and pain interference at 22 ± 2, 46 ± 2 and 70 ± 2 hours after the first dose.

On Day 4, following evaluations will be performed:

1. Review of adverse events.
2. Review of concomitant medications.
3. Blood draw (8 ± 3 mL) for assessment of SDE, nalbuphine, acetaminophen and metabolites (AAP-Sul, AAP-Glc, AAP-Cys, AAP-Nac and APAP-protein adducts) concentrations at 70.75 ± 2 hours after the first dose in all subjects and Blood draw (20 ± 3 mL) for CBC with differential, platelets and blood chemistry screen (Not include Antibody screening and ABO Grouping & RH Type determination). The blood collection time is carried out according to the routine blood drawing procedure in the hospital ward.
4. Physical examination, including vital signs and 12-lead ECG.
5. Patient satisfaction.
6. Galactose single-point (GSP) test.

Follow-up visit:

24 and 48 hours after the subject took the last medication then researchers conduct telephone interviews to track the overall condition of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≧ 20 years of age at Screening.
* Knee replacement patients.
* American Society of Anesthesiology Physical Class 1 and 2.
* Ability and willingness to provide informed consent, adhere to the study visit schedule and complete all study assessments and language specific questionnaires.

Exclusion Criteria:

* Body weight less than 50 kg.
* Subject is pregnant or breastfeeding. Women of childbearing potential have a positive urine pregnancy test at baseline.
* Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study.
* History of hypersensitivity or allergy to amide-type local anesthetics, opioid, acetaminophen, or any ingredient of the medications administered in this study.
* Subject has a resting respiratory rate less than 8 per minute and blood oxygen saturation less than 90 %.
* Administration of an investigational drug within 5 elimination half-lives of such investigational drug prior to study drug administration.
* The investigator judged that any psychiatric disorder or psychological condition that may interfere with study assessments or compliance.
* History of abuse illicit medications, prescription medicines or alcohol within the past 2 years. History or presence of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (the equivalent of 14 glasses of 120 mL wine or 14 cans of 350 mL beer).
* Current painful physical condition other than knee pain.
* The investigator judged that the sensory nerve examination results were abnormal before the knee replacement in this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of visual analogue scale | 0 hour - 70 hours after first dose
  Pain assessment calculated as the area under the curve (AUC) of visual analogue scale (VAS, 0-100 mm) pain intensity scores through 70 ± 2 hours after the first dose.

SECONDARY OUTCOMES:
The first time using any one kind of rescue medication | Day 1 - Day 4
  1. The first time using any one kind of rescue medication, in which the first-line rescue medication parecoxib 40 mg and second-line rescue medication morphine 4 mg.
Consumption of rescued parecoxib | Day 1 - Day 4
  2. Consumption of rescued parecoxib 40 mg and morphine 4 mg.
Brief Pain Inventory short form (BPIsf) | Day 2 - Day 4
  3. Using Brief Pain Inventory short form (BPIsf) to assess pain intensity and pain interference at 22 ± 0.5, 46 ± 0.5 and 70 ± 0.5 hours after the first dose.
The evaluation of adverse events | Day 1 - Day 6
  4. The evaluation of the number and frequency of adverse events will continue until the end of the trial 120 hours after the first dose.
Patient satisfaction | Day 4
  5. Patient satisfaction on day 4.
Assessment of ALT and AST | Day 4
  6. Assessment of ALT and AST at 70.75 ± 2 hours after the first dose.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Fong Mr Chen, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan